CLINICAL TRIAL: NCT03058224
Title: Randomized, Double-blind, Placebo-controlled Exploratory Trial to Investigate Efficacy and Safety of IGN-ES001 in Patients With Chronic Widespread Pain With or Without Fibromyalgia
Brief Title: Efficacy and Safety of IGN-ES001 in Chronic Widespread Pain With or Without Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IgNova GmbH (Industry)
Collaborators: Scope International AG (Industry); Klinar CRO (Other); CenTrial GmbH (Industry); Pharmasolutions4U (Unknown); idv Data Analysis and Study Planning (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IGN-ES001-CR01
Record Dates: First submitted 2017-02-09; First posted 2017-02-20 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Chronic Widespread Pain; Fibromyalgia
Keywords: Pain, Symptom Severity; Immunoglobulin IgY; Fibromyalgia; Widespread Pain Index; Eggyolk; FIQ-R; SF-36v2TM; MOS-SS; FSS; PGIC; Quality of life
MeSH Terms: conditions — Chronic Pain; Fibromyalgia; Pain | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IGN-ES001 (Experimental): Polyclonal avian immunoglobulin IgY containing specific IgY against E. coli F18ab and S. typhimurium in partially delipidated avian egg yolk powder
  Interventions: Drug: IGN-ES001; Drug: Parol 500 mg Tablets (acetaminophen)
- Placebo (Placebo Comparator): Polyclonal avian immunoglobulin IgY containing unspecific IgY in partially delipidated avian egg yolk powder
  Interventions: Drug: Parol 500 mg Tablets (acetaminophen)

INTERVENTIONS:
Drug: IGN-ES001 — Only active product will be compared with placebo as described in Arms and Interventions.
  Arms: IGN-ES001
Drug: Parol 500 mg Tablets (acetaminophen) — Analgesic Rescue Medication

SUMMARY:
This is a randomized, double-blind, placebo-controlled exploratory trial to investigate efficacy and safety of food supplement IGN-ES001 in patients with chronic widespread pain (CWP) with or without fibromyalgia (FM).

DETAILED DESCRIPTION:
Patients will perform five scheduled on-site visits and five phone calls:

* Screening visit, V1 (Day -10 to -7), informed consent
* Baseline visit, V2 (Day 1), randomization, treatment start
* Phone call, V3 (Day 4 ± 1)
* Phone call, V4 (Day 8 ± 3)
* Phone call, V5 (Day 15 ± 3)
* On-site visit, V6 (Day 22 ± 3)
* Phone call, V7 (Day 29 ± 3)
* Phone call, V8 (Day 36 ± 3)
* On-site visit, V9 (Day 43 + 3), treatment end
* Follow-up on-site visit, V10 (Day 50 + 7, or 7 + 7 days after EDV).

In addition, patients may be asked to return to the trial site between scheduled visits for assessment of safety data (unscheduled visits).

The maximum duration of treatment for the individual patient will be 46 days (including allowed visit window deviation). The maximum duration of trial participation for the individual patient will be 67 days.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female out-patient ≥ 18 years and ≤ 70 years of age.
2. Patient willing and able (e.g. mental and physical condition) to participate in all aspects of the trial, including use of investigational product, subjective completion of diaries and questionnaires, attending scheduled visits, completing telephone interviews, and compliant with protocol requirements as evidenced by providing signed writteninformed consent.
3. History of chronic widespread pain (for at least three months prior to visit V1 (screening)).
4. a.) For FM patients: Widespread Pain Index (WPI) ≥ 7 and Symptom Severity (SS) ≥ 5 or WPI 3-6 and SS ≥ 9 (original preliminary fibromyalgia criteria of the American College of Rheumatology (ACR) 2010).

   b.) For non-FM CWP patients: WPI ≥ 3-6 and SS ≥ 5-8 (modified from the preliminary fibromyalgia criteria of the ACR 2010).
5. Use of prior and concomitant medications/ therapies (if not excluded, see exclusion criteria no 6 and no 7), non-pharmacological therapies and lifestyle habits (e.g. diet changes, Ramadan participation, etc.) that could influence the efficacy assessments must have been stable for at least 30 days prior to visit V1 (screening) and are anticipated to be at a stable regimen throughout the trial until visit V9.
6. Patient has negative urine test at screening visit V1 for the following drugs of abuse:

   1. Amphetamine
   2. Cocaine
   3. Metamphetamine
   4. Morphine
   5. Tetrahydrocannabinol
7. Female patient is surgically sterile (i.e. bilateral tubal ligation, bilateral oophorectomy, or hysterectomy), or at least two years postmenopausal or, if of childbearing potential, she is sexually abstinent or agrees to practice adequate contraceptive measures (hormonal contraceptives, intrauterine device, double-barrier method).
8. Patient must have completed at least 6 screening phase diary pages satisfactorily within the past 7 days before visit V2.
9. Median pain NRS must be ≥ 4 in at least 1 out of the 6 pain qualities and ≥ 4 in overall pain assessment. The median will be calculated from the last 7 days before visit V2 (baseline) and will serve as baseline value.

If all inclusion criteria are fulfilled (and none of the exclusion criteria below), the patient will be randomized at visit V2 and continues in the trial. Otherwise the patient will be excluded from trial participation.

Exclusion Criteria:

1. Patients without a basic and stable CWP therapy which started at least 30 days before V1 (screening) i.e. treatment-naive patients, first diagnosis.
2. Known allergy or intolerance to egg or egg constituents.
3. History of or currently active malignancy except for malignancies that were successfully treated and have had no recurrence within 5 years before screening visit V1.
4. Known, uncontrolled endocrine disorders, such as hypothyroidism (TSH and free T4), and diabetes mellitus (HbA1c).
5. Known severe hepatic, renal, respiratory, hematologic, neurologic, infectious, or immunologic disease, unstable cardiovascular disease, or any other medical or psychiatric condition that, in the judgment of the investigator, would make the patient inappropriate for participation in this trial.
6. Immune response modulating medication/ therapy e.g. systemic corticosteroids, antibodies other than IP (investigational product) from a period starting 90 days before visit V1 (screening).
7. WHO step-II and step-III opioids (except occasional use of codeine as cough medication) from a period starting 60 days before visit V1 (screening).
8. Intractable vomiting likely to significantly influence gastrointestinal (GI) investigational product presence.
9. Surgery within 60 days before visit V1 (screening) or anticipated or scheduled for the next nine weeks after visit V1 (screening).
10. Vaccination from a period starting 30 days prior to visit V1 (screening).
11. Known liver disease or evidence of impaired hepatic function (total bilirubin, aspartate aminotransferase [ASAT], alanine transaminase [ALAT], gamma-glutamyltransferase [GGT], or alkaline phosphatase [AP] > 3 times the upper limit of normal).
12. Known kidney disease or evidence of impaired renal function, i.e. estimated glomerular filtration rate (eGFR) based on serum creatinine < 60 mL/min as calculated by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula.
13. Pregnancy or breastfeeding.
14. Known severe psychiatric illness (e.g. schizophrenia, major depression, anxiety disorder, obsessive compulsive disorder, panic disorder, social phobia, post-traumatic stress) or personality disorder (e.g. borderline personality). Obvious suicide risk.
15. Current and/ or history of known or suspected drug or substance abuse including alcohol abuse within five years before visit V1 (screening) as stated by the patient and/ or withdrawal symptoms.
16. Previous enrolment in this trial, or participation in any other studies involving investigational products, simultaneously or within six months prior to be screened for this trial (visit V1).
17. Persons committed to an institution by virtue of an order issued either by the judicial or other authorities.
18. Employee of the investigator or trial site, with direct involvement in the proposed trial or other studies under the direction of that investigator or trial site, as well as family members of the employees or the investigators.
19. Patients unable or unwilling to include yoghurt or ayran into their daily diet.
20. Severe diarrhea.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2017-02-16 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-12-08 (Actual)

PRIMARY OUTCOMES:
Pain, final percent changes from baseline (based on diary), univariate analysis | Six Weeks
  The overall pain improvement will be assessed by means of the percent changes from baseline (Visit 2) to end of treatment visit (Visit 9). Percent changes are preferred to raw changes due to their implicit adjustment for baseline differences in the case of proportional decrease. The baseline pain value will be calculated as mean overall pain of the last seven-day time period of the screening phase from Day -7 to Day -1. Minimum the last 6 out of 7 days prior to baseline visit V2 must be documented. The final pain value will be calculated as mean overall pain of the last seven-day time period prior to the end of the adjunctive treatment period from Day 36 to Day 42.
Pain, final percent changes from baseline (based on diary), multivariate analysis | Six Weeks
  In addition to the univariate analysis of the overall pain score, a correlation-sensitive multidimensional approach will be performed with respect to the two major pain activity levels:
  * Pain at rest (sum score of three locations), percent change from baseline
  * Pain perceived during physical strain (sum score of three locations), percent change from baseline
Pain, final responder (based on diary) | Six Weeks
  Responders will be defined as patients with a percent decrease from baseline of the overall pain score by at least 30%. This is a recommended benchmark for a "clinically meaningful improvement" (Farrar et al.), and provides robustness in case of proportional pain decrease (independency from baseline pain level). Tubach et al. (2012) defined a percent decrease of 20% as minimal clinically important change. Thus, the recommendation of Farrar et al. is regarded as optimum choice for a clinically meaningful responder definition.

SECONDARY OUTCOMES:
Responder* rate, alternative definition (based on diary) | Six Weeks
Change in Fibromyalgia Impact Questionnaire Revised version (FIQ-R) score from baseline (visit V2) | Six Weeks
Change in Short-Form-36 version 2 Quality-of-Life questionnaire (SF-36v2TM) score from baseline (visit V2) | Six Weeks
Change in Medical Outcomes Study Sleep Scale (MOS-SS) score from baseline (visit V2) | Six Weeks
Change in Fatigue Severity Scale (FSS) score from baseline (visit V2) | Six Weeks
Patient's Global Impression of Change (PCIG) Questionnaire | Six Weeks
  "The patients will rate their change in the overall status "since the start of the study, my overall status is" on a scale ranging from 1 (= very much improved) to 7 (= very much worse). Patients will complete the PGIC questionnaire at visit 9 (or at Early Discontinuation Visit) covering the whole 6-week treatment period from baseline visit 2."
Consumption of rescue medication | Six Weeks
Time to first rescue medication (days) | Dependent to the timeframe of the first rescue medication from first investigational product intake following baseline visit 2 through study completion, an average of six weeks

CONTACTS AND LOCATIONS:
Locations (23):
- Turkey (Türkiye) (23):
  - Çukurova University School of Medicine, Adana
  - Akdeniz University School of Medicine, Antalya
  - Adnan Menderes University School of Medicine, Aydin
  - Uludağ University School of Medicine, Bursa
  - Onsekiz Mart University School of Medicine, Çanakkale
  - Trakya University School of Medicine, Edirne
  - Gaziantep University School of Medicine, Gaziantep
  - Bezmialem Vakıf University School of Medicine, Istanbul
  - İstanbul Physical Treatment and Rehabilitation Training and Research Hospital, Istanbul
  - İstanbul University Cerrahpaşa School of Medicine, Istanbul
  - İstanbul University İstanbul School of Medicine, Istanbul
  - Maltepe University School of Medicine, Istanbul
  - Marmara University Pendik Training and Research Hospital, Istanbul
  - Şişli Florence Nighingale Hospital, Istanbul
  - Şişli Hamidiye Etfal Training and Research Hospital, Istanbul
  - İzmir Medical Park Hospital, Izmir
  - Erciyes UNiversity School of Medicine, Kayseri
  - Necmettin Erbakan University School of Medicine, Konya
  - Sakarya University School Of Medicine Korucuk Training and Research Hospital, Sakarya
  - Cumhuriyet University School of Medicine, Sivas
  - Namık Kemal University School of Medicine, Tekirdağ
  - Karadeniz Technical University School of Medicine, Trabzon
  - Bülent Ecevit University School of Medicine, Zonguldak

IPD SHARING:
Plan to Share IPD: No